CLINICAL TRIAL: NCT05072236
Title: Effects of Adding Intravenous Lidocaine, Alfentanil Before Bronchoscopic Insertion for Preventing Cough During Bronchoscopic Spraying of Local Anesthetics in Non-intubated Bronchoscoopic Interventions
Brief Title: Effects of Adding Different Drugs for Preventing Cough Induced by Bronchoscopic Spraying of Local Anesthetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 202107071MIND
Record Dates: First submitted 2021-09-14; First posted 2021-10-08 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-09

CONDITIONS: Lung Diseases; Total Intravenous Anesthesia; Bronchoscopic Interventions
Keywords: cough; desaturation; ventilation; bronchoscopic interventions
MeSH Terms: conditions — Lung Diseases; Cough; Respiratory Aspiration | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- normal saline (Placebo Comparator): intravenous normal saline 5 mL 1 minute before bronchoscope insertion
  Interventions: Procedure: bronchoscopic insertion
- lidocaine (Active Comparator): intravenous lidocaine 1.5 mg/kg 1 minute before bronchoscope insertion
  Interventions: Procedure: bronchoscopic insertion
- alfentanil (Experimental): intravenous alfentanil 10 ug/kg 1 minute before bronchoscope insertion
  Interventions: Procedure: bronchoscopic insertion

INTERVENTIONS:
Procedure: bronchoscopic insertion — After intravenous anesthesia is stabilized with BIS levels between 50-70, Intravenous lidocaine 1.5 mg/kg, or alfentanil 10 ug/kg, or 5 mL normal saline will be injected. Bronchoscopic insertion will be started 1 minute later. After seeing the vocal cords, local spraying of 2% will be initiated from vocal cords, trachea, and bilateral bronchial trees.
  Other Names: bronchoscopic spraying of 2% lidocaine

SUMMARY:
Cough is the most unwanted response during bronchoscopic interventions for hemodynamic instability, hypoxemia, and interruption of interventions. Topical lidocaine is recommended with a grade evidence in British Thoracic Society guideline. However, severe cough often induces during the initial bronchoscopic spraying of local anesthesia, follows with uneven spraying, spasm or arrythmias. In previous reports, there were many drugs and techniques investigated for preventing cough during broncoscopic spraying. As bronchoscopic interventions need more space and stability of airways to precisely operate on, few studies have focused on the effects of different drugs for preventing cough. In this study, Different intravenous drugs (lidocaine, alfentanil, compared to normal saline) is planned to be injected one minutes before bronchoscopic insertion, the responses to bronchoscopicly spraying local anestheticsuch as cough intensity, BIS levels, ANI, Transdermal O2 and CO2, respiration were recorded and analyzed.

DETAILED DESCRIPTION:
Cough is the most unwanted response during bronchoscopic interventions. Cough could lead to airway spasm, hemodynamic instability, desaturation, hypoventilation, and then interrupt the following interventions. In previous reports, lodicaine and other drugs given intravenously, inhalationally or trans-cricoidally have been investigated for preventing cough during conventional broncoscopic examinations. As bronchoscopic interventions were goaled to precise localization and operations with higher yield rate. Steady airways without endotracheal tubes are usually required. Topical lidocaine is recommended with a grade evidence in British Thoracic Society guideline. However, severe cough often induces during the initial bronchoscopic spraying of local anesthesia, follows with uneven spraying, spasm or arrythmias. There are few studies focused on the effects of different drugs for preventing cough even bronchoscopic spary of local anesthetics has become the routine pratice before interventions. In this study, different intravenous drugs (lidocaine, alfentanil, compared to normal saline) are planned to be injected one minutes before bronchoscopic insertion, the responses to bronchoscopic spraying local anesthetic were recorded and analyzed. Besdies cough scores, the following changes are recorded and compared: (1) status on visualization and the responses to spraying of vocal cords, (2) anesthetic depth (BIS levels), ANI scores (3) blood pressure and heart beats, (4) data of hemoglobin saturation (SPO2) and Transdermal O2 and CO2. We goaled to compare the effects of intravenous lidocaine and etomidate on cough intensity, hemodynamics, ventilation, and bronchoscopic withdrawl rate during bronchoscopic interventions with intravenous anethesia.

ELIGIBILITY:
Inclusion Criteria:

* patients planned to receive bronchoscopic interventions for lung tumors with intravenous anesthesia.

Exclusion Criteria:

* conventional bronchoscopy without interventions such as EBUS, tracheal tumore excision

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
cough score | from bronchoscopic spray local anesthetics on vocal cords to the end of spraying on bonchial trees
  cough severity x times Cough severity was graded on a 5-point scale: minimal cough, 1 point; moderate cough, 2 points; severe cough, 3 points; bouts of coughing, 4 points; and series of bouts of coughing, 5 points.
BIS levels from EEG monitor | from 1 minutes before bronchoscopic insertion to 20 minutes after bronchoscopic interventions
  the changes of BIS levels (0-100)
ANI scores from analgesia-nociception monitor (0-100) | from 1 minutes before bronchoscopic insertion to 20 minutes after bronchoscopic interventions
  the changes of ANI scores (0-100)

SECONDARY OUTCOMES:
MAP | from bronchoscopic insertion to 20 minutes after completion of local anesthetic spraying
  mean arterial pressure, mmHg
heart rate | from bronchoscopic insertion to 20 minutes after completion of local anesthetic spraying
  heart rate, beats/ minute
SPO2 | from bronchoscopic insertion to 20 minutes after completion of local anesthetic spraying
  SPO2, %
Transdermal CO2 | from bronchoscopic insertion to 20 minutes after completion of local anesthetic spraying
  Transdermal CO2, mmHg
BTransdermal O2 | from bronchoscopic insertion to 20 minutes after completion of local anesthetic spraying
  Transdermal O2, mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Yajung Cheng, Study Chair — National Taiwan University Hospital, Cancer Center
Locations (1):
- National Taiwan University Cancer Center Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No